CLINICAL TRIAL: NCT07310498
Title: The Effects of 10-week Complex Training on Physical Characteristics, Biomechanics and Fitness of Chinese National Korfball Players.
Brief Title: 10-week Complex Training for Chinese National Korfball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/KK/23110824
Record Dates: First submitted 2025-09-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Plyometric Exercises; Fitness Training; Athlete; Physical Fitness; Biomechanical Data; Athletic Performance

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by sex into two equally sized groups (male and female). Both groups will receive the same 10-week unilateral complex training intervention. No between-group comparisons are planned; analyses will focus on within-group pre- to post-intervention changes.
Masking Description: This is an open-label study; both participants and investigators are aware of the intervention being administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 10-week Unilateral Complex Training (Experimental): Participants will be stratified by sex into two equally sized groups (male and female). All participants will complete the same 10-week unilateral complex training program, which combines resistance and plyometric exercises within each session. No between-group comparisons are planned; analyses will focus on pre- to post-intervention changes.
  Interventions: Behavioral: 10-week Unilateral Complex Training Program

INTERVENTIONS:
Behavioral: 10-week Unilateral Complex Training Program — Participants will undergo a 10-week unilateral complex training program. Each training session combines resistance exercises (e.g., squats, lunges, or weighted lower-limb movements) with plyometric exercises (e.g., jumps, bounding, or explosive step-back movements) performed in alternating sequence. Training is delivered three times per week under supervision. All participants, divided equally by sex, follow the same program. The intervention is designed to improve strength, power, balance, and shooting performance while reducing interlimb asymmetry. No between-group comparisons are planned; outcomes are assessed pre- and post-intervention.

SUMMARY:
Korfball is a mixed-gender team sport that requires high levels of coordination, balance, and physical fitness. Unlike basketball or netball, players cannot dribble or run with the ball, and shots must often be taken in a single-leg, step-back position. These unique demands create challenges for athletes' strength, balance, and injury prevention. Despite korfball's growing popularity, scientific research on the sport's physical, biomechanical, and training characteristics remains limited.

Complex training (CT) is a training method that alternates heavy resistance exercises with plyometric movements. This approach is known to improve strength, power, sprinting, and jumping ability in other team sports. It is especially relevant for unilateral sports movements, which are common in korfball shooting and defensive actions. However, no studies to date have applied CT to korfball athletes, and the effects of such training on their performance, biomechanics, and interlimb asymmetries are unclear.

This study is designed to address three research areas:

To describe the internal and external load characteristics of korfball matches using heart rate monitoring and video-based analysis.

To investigate limb asymmetry in korfball players through assessments of biomechanics, anthropometry, physical fitness, and shooting technique.

To evaluate whether a 10-week unilateral complex training program can reduce limb asymmetry and improve physical fitness and shooting performance in elite players.

The study includes both cross-sectional and interventional components. First, competition loads will be monitored to understand game-specific demands. Second, assessments will compare dominant and non-dominant limbs in terms of strength, biomechanics, and technical performance. Finally, athletes will undergo a 10-week unilateral complex training program, after which the same measures will be repeated to test for improvements.

The expected outcomes are a clearer understanding of the physiological and biomechanical characteristics of korfball players, as well as evidence on the effectiveness of unilateral complex training. This knowledge may guide coaches and practitioners in designing targeted training strategies to enhance performance, reduce injury risk, and optimize athlete development in korfball.

ELIGIBILITY:
Inclusion Criteria:

* Male or female athletes aged 18 to 35 years.
* Selected for the China National Korfball Team or the China Youth National Korfball Team.
* Able to participate in the full training and testing protocol and willing to provide informed consent.

Exclusion Criteria:

* Participation in structured physical training other than korfball training within the previous 6 months.
* History of cruciate ligament injury, fracture, or other significant injury affecting sports performance within the previous 12 months.
* Failed routine musculoskeletal health screening or has unresolved injury/medical condition that precludes safe participation.
* Does not meet baseline strength prerequisites required for safe participation in complex training (combined resistance and plyometric exercises) according to NSCA guidelines.

Additional notes (for study procedures, not eligibility):

-Participants will complete an information questionnaire to document training history and basic characteristics.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 10 in 1-Repetition Maximum (1RM) Back Squat (kg) | Baseline and Week 10
  Maximal lower-body strength assessed as the one-repetition maximum (1RM) load for the barbell back squat. Participants completed standardized warm-up sets followed by progressive single attempts to determine the maximal load successfully lifted once with correct technique; rest periods were provided between attempts. The outcome is the 1RM load, reported in kilograms (kg).

SECONDARY OUTCOMES:
1-Repetition Maximum (1RM) Shoulder Press (kg) | Baseline and Week 10
  Upper-body maximal strength assessed as the one-repetition maximum (1RM) load for the shoulder press exercise. The 1RM is defined as the maximal load that can be lifted once with correct technique for the specified exercise; the outcome is the 1RM load, reported in kilograms (kg).
Y-Balance Test Composite Score (percent) | Baseline and Week 10
  Dynamic balance assessed using the Lower Quarter Y-Balance Test. Composite score calculated as ((ANT + PM + PL) / (3 × limb length)) × 100; reported as percent.
Single-Leg Triple Hops (m) | Baseline and Week 10
  Single-leg triple hop for distance and reported in meters（m）.
Yo-Yo Intermittent Recovery Test Total Distance (m) | Baseline and Week 10
  Intermittent running performance assessed using the Yo-Yo Intermittent Recovery Test Level 1 (YYIR1). Performance is defined as the maximal total distance completed, reported in meters (m).
T-Test Agility Time (s) | Baseline and Week 10
  Agility assessed using the T-test; outcome is time to complete the course, reported in seconds (s).
Isokinetic Hip Extension Peak Torque/Body Mass at 60°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for hip extension measured using an isokinetic dynamometer at 60°/s; normalized to body mass and reported as N·m/kg.
Isokinetic Hip Extension Peak Torque/Body Mass at 180°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for hip extension measured using an isokinetic dynamometer at 180°/s; normalized to body mass and reported as N·m/kg.
Isokinetic Knee Extension Peak Torque/Body Mass at 60°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for knee extension measured using an isokinetic dynamometer at 60°/s; normalized to body mass and reported as N·m/kg.
Isokinetic Knee Extension Peak Torque/Body Mass at 180°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for knee flexion measured using an isokinetic dynamometer at 180°/s; normalized to body mass and reported as N·m/kg.
Isokinetic Ankle Extension (Plantarflexion) Peak Torque/Body Mass at 60°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for ankle extension (plantarflexion) measured using an isokinetic dynamometer at 60°/s; normalized to body mass and reported as N·m/kg.
Isokinetic Ankle Extension (Plantarflexion) Peak Torque/Body Mass at 180°/s (N·m/kg) | Baseline and Week 10
  Concentric peak torque for ankle extension (plantarflexion) measured using an isokinetic dynamometer at 180°/s; normalized to body mass and reported as N·m/kg.
Step-back Jump Shot Vertical Impulse (N·s/kg) | Baseline and Week 10
  Vertical GRF impulse (Z-axis) during the propulsion phase of the step-back jump shot, computed as the time integral of the Z-axis GRF over propulsion and normalized to body mass (N·s/kg). Registered value = bilateral mean; limb-specific (left/right) values will be reported as additional analyses.
Step-back Jump Shot Jump Height (cm) | Baseline and Week 10
  Jump height during the step-back jump shot will be derived from force-plate-defined flight time and reported in centimeters (cm). The registered outcome value will be the bilateral mean; limb-specific values will be reported as additional analyses.
Squat Jump Height (cm) | Baseline and Week 10
  Squat jump height derived from force plate data (flight-time method ) and reported in centimeters (cm). Registered value = bilateral mean; limb-specific values reported as additional analyses.
Drop Jump Reactive Strength Index (RSI) (m/s) | Baseline and Week 10
  Reactive Strength Index (RSI) during drop jump, calculated as jump height (m) divided by ground contact time (s); reported as m/s. Registered value = bilateral mean; limb-specific values reported as additional analyses.
Change-of-Direction (45°) Braking Impulse (N·s/kg) | Baseline and Week 10
  Braking GRF impulse in the sagittal axis (Y-axis) during the 45° change-of-direction task, computed as the time integral of the braking-direction portion of the Y-axis GRF over the braking/weight-acceptance interval (initial contact to peak knee flexion) and normalized to body mass (N·s/kg). The registered outcome value will be the bilateral mean; limb-specific values (left/right) will be reported as additional analyses.
Change from Baseline to Week 10 in Overall Shooting Accuracy Across 3 m, 5 m, and 7 m in a 1-Minute Timed Shooting Protocol (%) | Baseline and Week 10
  Shooting accuracy will be assessed using a standardized sport-specific timed shooting protocol at three distances (3 m, 5 m, 7 m). At each distance, participants will attempt as many shots as possible within 1 minute. The number of successful shots and total shot attempts will be recorded at each distance. The registered outcome value will be overall shooting accuracy (%) aggregated across all three distances, calculated as: (total successful shots across 3 m+5 m+7 m ÷ total shot attempts across 3 m+5 m+7 m) × 100. Distance-specific accuracies (3 m, 5 m, 7 m) will be analyzed and reported as additional analyses.

OTHER OUTCOMES:
Body Mass Index (BMI) (kg/m²) | Baseline and Week 10
  BMI will be calculated as body mass in kilograms divided by the square of stature in meters and reported as kg/m².
Body Fat Percentage (%) | Baseline and Week 10
  Body fat percentage will be assessed using a bioelectrical impedance analysis (BIA) body composition analyzer under standardized conditions. Results will be recorded as percent (%).
Mid-thigh Girth (cm) | Baseline and Week 10
  Mid-thigh girth will be measured with a non-elastic tape at the midpoint between the inguinal crease and the proximal border of the patella, perpendicular to the long axis of the thigh, and recorded in centimeters (cm).
Maximal Calf Girth (cm) | Baseline and Week 10
  Maximal calf girth will be measured with a non-elastic tape at the level of the largest calf circumference and recorded in centimeters (cm).
Change from Baseline to Week 10 in Limb Symmetry Index (LSI) for Isokinetic Muscle Strength Test in 180° (%) | Baseline and Week 10
  LSI will be calculated for concentric knee extension peak torque at 180°/s as: LSI = (dominant limb / non-dominant limb) × 100, reported as percent (%). Peak torque will be normalized to body mass (N·m/kg) before LSI calculation. Dominant limb defined a priori.
Change from Baseline to Week 10 in Drop Jump RSI LSI (%) | Baseline and Week 10
  LSI will be calculated for drop jump Reactive Strength Index (RSI) as: LSI = (dominant limb / non-dominant limb) × 100, reported as percent (%). RSI will be computed as jump height (m) divided by ground contact time (s) for each limb. Dominant limb will be defined a priori.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Sport University, Zhenzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR